CLINICAL TRIAL: NCT06215586
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Clinical Study to Assess the Safety and Effectiveness of Tovinontrine in Patients With Chronic Heart Failure With Preserved Ejection Fraction
Brief Title: Safety & Effectiveness of Tovinontrine in Chronic Heart Failure With Preserved Ejection Fraction (Cycle-2-PEF)
Acronym: Cycle-2-PEF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cardurion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRD-750-202; 2023-508737-13 (EudraCT Number)
Record Dates: First submitted 2023-12-13; First posted 2024-01-22 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure; Heart Failure Preserved Ejection Fraction; Cardiovascular Diseases; Heart Diseases
Keywords: PDE9; PED9 Inhibitor; Heart Failure; CRD-750; Tovinontrine; HFpEF
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tovinontrine (CRD-750) (Experimental)
  Interventions: Drug: Tovinontrine (CRD-750
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tovinontrine (CRD-750 — Tablets administered orally
  Arms: Tovinontrine (CRD-750)
Drug: Placebo — Tablets administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of tovinontrine compared to placebo to lower NT-proBNP in patients with chronic heart failure with preserved ejection fraction

ELIGIBILITY:
Inclusion Criteria:

* Is an adult male or female patient ≥ 18 years of age
* Has evidence in the medical history supporting a diagnosis of clinical HF syndrome, NYHA functional class II to III, with the duration of at least 6 months prior to the time of Screening. The HF syndrome is defined by documentation of 1 or more of the following:

  * At least 1 of the typical symptoms due to HF such as dyspnea and/or fatigue limiting exercise capacity;
  * At least 1 of the typical signs of HF such as peripheral edema, elevated jugular venous pressure, pulmonary crackles; or
  * Hospitalization, emergency department visit, or outpatient visit for HF requiring intravenous (IV) or subcutaneous (SQ) diuresis within the past 12 months.
* Has ejection fraction (EF) >40% and left atrial enlargement by transthoracic echocardiogram (TTE) performed and interpreted locally at the time of Screening;
* Has NT-proBNP level ≥ 300 pg/mL at the time of Screening. Patients with atrial fibrillation or flutter at the time of Screening are required to have an NT proBNP level of ≥500 pg/mL at the time of Screening;
* Is on stable optimized doses of guideline-directed HF therapy, per Investigator's clinical judgment, for a minimum of 4 weeks prior to the time of Screening and during the Screening Period, with no planned changes after randomization; Has had no addition of new guideline-directed HF therapy within the 3 months prior to the time of Screening or during the Screening Period;

Exclusion Criteria:

* Has documented EF ≥ 60% by TTE within 6 months of the time of Screening or during the Screening Period;
* Has evidence of recent HF exacerbation defined by hospitalization or requirement for IV or SQ diuretics within 60 days of the time of Screening or during the Screening Period;
* Has a requirement for routine, scheduled outpatient IV infusions for HF (ie, inotropes, vasodilators, or diuretics) or routinely scheduled ultrafiltration;
* Has elective interventions (eg, percutaneous coronary intervention, device implantations, percutaneous structural heart disease interventions, cardiac and non-cardiac surgery) planned to occur during involvement in this study;
* Has acute coronary syndrome, stroke, transient ischemic attack, cardiac, carotid or other major cardiovascular surgery, or carotid angioplasty within 60 days of the time of Screening or during the Screening Period;
* Has had a prior or planned orthotopic heart transplantation;
* Has presence of or plan for mechanical circulatory support;

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2024-02-13 (Actual); Primary Completion 2025-09-02 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
Change in biomarkers from Baseline to Week 12 - NT-proBNP | Baseline to Week 12
  The percent change in plasma NT-proBNP from Baseline to Week 12.

SECONDARY OUTCOMES:
Change in biomarkers at week 12 by treatment group - cGMP | Baseline to Week 12
  The percent change in urine and plasma cGMP from Baseline to Week 12.
Change in biomarkers at week 12 by treatment group - BNP | Baseline to Week 12
  The percent change in BNP from Baseline to Week 12.
Change in the biomarker ratio at Week 12 - NT-proBNP | Baseline to Week 12
  The percent change in the urine and plasma cGMP to NT-proBNP ratio at week 12.
Change in the biomarker ratio at Week 12 - BNP | Baseline to Week 12
  The percent change in the urine and plasma cGMP to BNP ratio from Baseline to Week 12.
The change from baseline in the Kansas City Cardiomyopathy Questionnaire-23 (KCCQ-23) | Baseline to Week 12
  Scaled 0 to 100 where lower scores represent worse health status than higher scores
The change from baseline in the KCCQ-23-CSS | Baseline to Week 12
  The proportion of patients with a ≥5, 10, and 20-point improvement in the KCCQ-23-CSS at Week 12
New York Heart Association (NYHA) classification at Week 12 | Week 12
  The post-baseline NYHA classification at Week 12
Treatment Emergent Adverse Events (TEAEs) | Baseline to Week 12
  The number of participants with TEAEs including drug related AEs, serious AEs (SAEs), and AEs leading to study drug discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Gail Berman, Study Director — Senior VP Head, Clinical Development Cardurion
Locations (80):
- United States (22):
  - Cardurion Investigative Site, Birmingham, Alabama
  - Cardurion Investigative Site, Little Rock, Arkansas
  - Cardurion Investigative Site, Orange, California
  - Cardurion Investigative Site, Torrance, California
  - Cardurion Investigative Site, Van Nuys, California
  - Cardurion Investigative Site, Jacksonville, Florida
  - Cardurion Investigative Site, Miami, Florida
  - Cardurion Investigative Site, Hazel Crest, Illinois
  - Cardurion Investigative Site, Peoria, Illinois
  - Cardurion Investigative Site, Alexandria, Louisiana
  - Cardurion Investigative Site, Covington, Louisiana
  - Cardurion Investigative Site, St Louis, Missouri
  - Cardurion Investigative Site, Buffalo, New York
  - Cardurion Investigative Site, New York, New York
  - Cardurion Investigative Site, Cleveland, Ohio
  - Cardurion Investigative Site, Oklahoma City, Oklahoma
  - Cardurion Investigative Site, Portland, Oregon
  - Cardurion Investigative Site, Rapid City, South Dakota
  - Cardurion Investigative Site, Nashville, Tennessee
  - Cardurion Investigative Site, Dallas, Texas
  - Cardurion Investigative Site, McKinney, Texas
  - Cardurion Investigative Site, Burlington, Vermont
- Cardurion Investigative Site, Chermside, Australia
- Belgium (2):
  - Cardurion Investigative Site, Bruges
  - Cardurion Investigative Site, Sint-Niklaas
- Bulgaria (6):
  - Cardurion Investigative Site, Burgas
  - Cardurion Investigative Site, Gabrovo
  - Cardurion Investigative Site, Plovdiv
  - Cardurion Investigative Site, Rousse
  - Cardurion Investigative Site, Sofia
  - Cardurion Investigative Site, Stara Zagora
- Canada (6):
  - Cardurion Investigative Site, Cambridge, Ontario
  - Cardurion Investigative Site, Hamilton, Ontario
  - Cardurion Investigative Site, Chicoutimi, Quebec
  - Cardurion Investigative Site, Montreal, Quebec
  - Cardurion Investigative Site, Sherbrooke, Quebec
  - Cardurion Investigative Site, Trois-Rivières, Quebec
- Czechia (2):
  - Cardurion Investigative Site, Hradec Králové
  - Cardurion Investigative Site, Prague
- Germany (5):
  - Cardurion Investigative Site, Elsterwerda, Brandenburg
  - Cardurion Investigative Site, Papenburg, Lower Saxony
  - Cardurion Investigative Site, Brandenburg, State of Berlin
  - Cardurion Investigational Site, Dresden
  - Cardurion Investigative Site, Magdeburg
- Hungary (5):
  - Cardurion Investigative Site, Balatonfüred
  - Cardurion Investigative Site, Budapest
  - Cardurion Investigative Site, Gyöngyös
  - Cardurion Investigative Site, Hatvan
  - Cardurion Investigative Site, Orosháza
- Cardurion Investigative Site, Milan, Italy
- Netherlands (5):
  - Cardurion Investigative Site, Eindhoven
  - Cardurion Investigative Site, Groningen
  - Cardurion Investigative Site, Hardenberg
  - Cardurion Investigative Site, Sneek
  - Cardurion Investigative Site, Zutphen
- Cardurion Investigative Site, Dunedin, New Zealand
- Poland (7):
  - Cardurion Investigative Site, Grodzisk Mazowiecki
  - Cardurion Investigative Site, Lodz
  - Cardurion Investigative Site, Lublin
  - Cardurion Investigative Site, Sopot
  - Cardurion Investigative Site, Torun
  - Cardurion Investigative Site, Warsaw
  - Cardurion Investigative Site, Wroclaw
- Spain (5):
  - Cardurion Investigative Site, Córdoba
  - Cardurion Investigative Site, Málaga
  - Cardurion Investigative Site, Santiago de Compostela
  - Cardurion Investigative Site, Seville
  - Cardurion Investigative Site, Valencia
- Taiwan (4):
  - Cardurion Investigative Site, Kaohsiung City
  - Cardurion Investigative Site, Taipei
  - Cardurion Investigative Site, Taipei County
  - Cardurion Investigative Site, Taoyuan District
- United Kingdom (8):
  - Cardurion Investigative Site, Bridgend
  - Cardurion Investigative Site, Chichester
  - Cardurion Investigative Site, Dundee
  - Cardurion Investigative Site, Glasgow
  - Cardurion Investigative Site, Harrow
  - Cardurion Investigative Site, Isleworth
  - Cardurion Investigative Site, London
  - Cardurion Investigative Site, Southampton

IPD SHARING:
Plan to Share IPD: No